CLINICAL TRIAL: NCT00862693
Title: Calcitriol in the Treatment of Immunoglobulin A Nephropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Renal Division, Peking University First Hospital, Key Laboratory of Renal Disease, Ministry of Health of China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20090315
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2009-03

CONDITIONS: Glomerulonephritis; Autoimmune Diseases
Keywords: Immunoglobulin A; Antibodies; treatment
MeSH Terms: conditions — Glomerulonephritis; Autoimmune Diseases | interventions — Calcitriol

ARMS (2):
- 1 calcitriol (Experimental): calcitriol 0.5ug/BIW for 12 months
  Interventions: Drug: Calcitriol
- 2 (No Intervention): no intervention

INTERVENTIONS:
Drug: Calcitriol — 0.5ug/Biw
  Arms: 1 calcitriol

SUMMARY:
Immunoglobulin A (IgA) nephropathy is the common primary glomerulonephritis in the world. Much literature suggests that vitamin D and its analogs have profound effects on immune system function and glomerular mesangial cell proliferation. Therefore, the investigators plan to conduct a randomized clinical study to evaluate the efficacy of Calcitriol in the treatment of IgA nephropathy. Forty patients with biopsy-proven IgA nephropathy will be recruited. They will be randomized to Calcitriol for six months or no treatment. Proteinuria, renal function, serum and urinary inflammatory markers will be monitored. This study will explore the potential anti-proteinuric and anti-inflammatory effects of Calcitriol in the treatment of IgA nephropathy, which has no specific treatment at present.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Biopsy-confirmed IgA nephropathy
* Proteinuria > 0.8 g/day in 3 consecutive samples within 12 weeks despite ACE inhibitor or angiotensin receptor blocker treatment for at least 3 months or estimated glomerular filtration rate < 60 ml/min/1.73m2
* Corrected serum calcium level < or = 2.45 mmol/l
* Willingness to give written consent and comply with the study protocol

Exclusion Criteria:

* Pregnancy, lactating or childbearing potential without effective method of birth control
* Severe gastrointestinal disorders that interfere with their ability to receive or absorb oral medication
* History of malignancy, including leukemia and lymphoma within the past 2 years
* Systemic infection requiring therapy at study entry
* Any other severe coexisting disease such as, but not limited to, chronic liver disease, myocardial infarction, cerebrovascular accident, malignant hypertension
* History of drug or alcohol abuse within past 2 years
* Participation in any previous trial on paricalcitol
* Patients receiving treatment of vitamin D and/or its analogue for other medical reasons within the past 3 months
* Patients receiving treatment of corticosteroid
* On other investigational drugs within last 30 days
* History of a psychological illness or condition such as to interfere with the patient's ability to understand the requirement of the study
* History of non-compliance
* Known history of sensitivity or allergy to paricalcitol or other vitamin D analogs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-08 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
decline of urine protein | 12 months treatment
  analysis urine protein after 12 months treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Renal Division, Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639